CLINICAL TRIAL: NCT00347074
Title: A Clinical Study of Keratoconus in Asian Patients and Assessment of Different Topographic Patterns of Keratoconus in Asian Patients
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R317/10/03
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2006-07-07 (Estimated); Status verified 2003-09

CONDITIONS: Keratoconus
Keywords: Keratoconus, corneal topography, ocular aberrometry, visual outcome, contact lens wear, quality of life
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
A clinical study of keratoconus in Asian Patients and assessment of different topographic patterns of keratoconus in Asian patients

DETAILED DESCRIPTION:
This hospital-based observational prospective study was designed to describe the characteristics of patients with keratoconus in an Asian population, Patients with keratoconus and keratoconus suspects presenting to the Singapore National Eye Centre who met the eligibility criteria are were recruited for this study. The following data were assessed:

1. Demographic characteristics of patients with keratoconus
2. Quality of life assessment in patients with keratoconus
3. Visual Outcome and management of keratoconus in terms of contact lens fitting
4. Corneal topographic patterns of patients with keratoconus
5. Aberrometry studies with regards to diagnosis of keratoconus and quality of vision in patients with keratoconus.

The patients not wearing contact lenses completed the study within one visit whereas the patients wearing contact lenses required 2 visits (one with contact lens wear and one without contact lens wear) to complete the study. For patients wearing contact lenses, they were advised to stop soft or rigid contact lens wear for 3 days before the initial visual acuity, subjective refraction, keratometry, Tomey and Orbscan II topography examinations and Wavefront aberrometry tests were performed.

Informed consent was obtained from all subjects after the nature of the study had been fully explained. The study gained approval from the Ethics Committee of the Singapore Eye Research Institute .

Each study participant was asked to answer the demography questionnaire form regarding their daily habit, medical history, economic and educational level and vision-related quality of life, and the Visual Function Index (VF-14).

Visual acuity was assessed in each eye using a logMAR chart. The visual acuity with manifest refraction was deemed the best corrected visual acuity(BCVA) for those patients who did not wear contact lenses, and the visual acuity with over-refraction (refraction over their contact lenses) for contact lens wearers.

Contrast sensitivity was examined only in patients with their habitual contact lenses in each eye using the Vision Contrast Test System (VCTS) chart (VCTS 6500 contrast sensitivity Chart) in 6 spatial frequencies.

Slit lamp evaluation and contact lens fit assessment were performed. Type of contact lens wear was recorded.

Corneal topography was performed using Tomey keratoconus screening system (Topographic Modeling System, software version 2.4.2J) without pupil dilation and without contact lens wear and the Orbscan II corneal topography system (Bausch &Lomb Surgical).

Ocular wavefront aberrations were measured across the central 6-mm dilated pupil (1% Tropicamide) of each eye with the Bausch and Lomb Technolas Zywave aberrometer with Zywave software version 4.45 (ZYOPTIX Diagnostic Workstation, Bausch & Lomb).

ELIGIBILITY:
Inclusion Criteria:

* Patients with keratoconus and keratoconus suspect presenting to the Singapore National Eye Centre who are willing to participate in the study

Exclusion Criteria:

* Patients with previous ocular surgery or trauma. Patients unwilling to participate in the study.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2003-09; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Li - Lim, FRCS(Ed), Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

REFERENCES:
- [Background] Krachmer JH, Feder RS, Belin MW. Keratoconus and related noninflammatory corneal thinning disorders. Surv Ophthalmol. 1984 Jan-Feb;28(4):293-322. doi: 10.1016/0039-6257(84)90094-8. PMID 6230745
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Maeda N, Klyce SD, Smolek MK. Comparison of methods for detecting keratoconus using videokeratography. Arch Ophthalmol. 1995 Jul;113(7):870-4. doi: 10.1001/archopht.1995.01100070044023. PMID 7605277
- [Background] Zadnik K, Barr JT, Edrington TB, Everett DF, Jameson M, McMahon TT, Shin JA, Sterling JL, Wagner H, Gordon MO. Baseline findings in the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study. Invest Ophthalmol Vis Sci. 1998 Dec;39(13):2537-46. PMID 9856763
- [Background] Rabinowitz YS. Videokeratographic indices to aid in screening for keratoconus. J Refract Surg. 1995 Sep-Oct;11(5):371-9. doi: 10.3928/1081-597X-19950901-14. No abstract available. PMID 8528916
- [Background] Maeda N, Klyce SD, Smolek MK, Thompson HW. Automated keratoconus screening with corneal topography analysis. Invest Ophthalmol Vis Sci. 1994 May;35(6):2749-57. PMID 8188468
- [Background] Smolek MK, Klyce SD. Current keratoconus detection methods compared with a neural network approach. Invest Ophthalmol Vis Sci. 1997 Oct;38(11):2290-9. PMID 9344352
- [Background] Rao SN, Raviv T, Majmudar PA, Epstein RJ. Role of Orbscan II in screening keratoconus suspects before refractive corneal surgery. Ophthalmology. 2002 Sep;109(9):1642-6. doi: 10.1016/s0161-6420(02)01121-1. PMID 12208710
- [Background] Pflugfelder SC, Liu Z, Feuer W, Verm A. Corneal thickness indices discriminate between keratoconus and contact lens-induced corneal thinning. Ophthalmology. 2002 Dec;109(12):2336-41. doi: 10.1016/s0161-6420(02)01276-9. PMID 12466180
- [Background] Maeda N, Fujikado T, Kuroda T, Mihashi T, Hirohara Y, Nishida K, Watanabe H, Tano Y. Wavefront aberrations measured with Hartmann-Shack sensor in patients with keratoconus. Ophthalmology. 2002 Nov;109(11):1996-2003. doi: 10.1016/s0161-6420(02)01279-4. PMID 12414405